CLINICAL TRIAL: NCT00093483
Title: Arsenic Trioxide, High-Dose Cytarabine and Idarubicin Induction Therapy in Previously Untreated de Novo and Secondary Adult Acute Myeloid Leukemia Patients < 60 Years Old - A Phase I Study
Brief Title: Arsenic Trioxide, Cytarabine, and Idarubicin in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000387999; P30CA016056 (NIH); RPCI-RP-0209
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Leukemia
Keywords: adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; untreated adult acute myeloid leukemia; secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Congenital Abnormalities | interventions — Filgrastim; Arsenic Trioxide; Cytarabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim — Subcutaneously beginning 12 hours after the last dose of chemotherapy and continuing until blood counts recover.
Drug: arsenic trioxide — IV over 1 hour on day 1
Drug: cytarabine — IV over 1 hour every 12 hours on days 1-6
Drug: idarubicin — IV over 30 minutes on days 2-4 (immediately after doses 3, 5 and 7 of cytarabine).

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as arsenic trioxide, cytarabine, and idarubicin, work in different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of arsenic trioxide when given together with cytarabine and idarubicin in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and/or biologically effective dose of arsenic trioxide followed by high-dose cytarabine and idarubicin in patients with previously untreated de novo or secondary acute myeloid leukemia.

OUTLINE: This is a dose-escalation study of arsenic trioxide. Patients are stratified according to timing of accrual (before November 2002 vs since November 2002).

Patients receive arsenic trioxide IV over 1 hour on day 1 followed by high-dose cytarabine IV over 1 hour every 12 hours on days 1-6 and idarubicin IV over 30 minutes on days 2-4 (immediately after doses 3, 5 and 7 of cytarabine). Patients also receive filgrastim (G-CSF) subcutaneously beginning 12 hours after the last dose of chemotherapy and continuing until blood counts recover.

Cohorts of 3-6 patients receive escalating doses of arsenic trioxide until the maximum tolerated dose (MTD), current dose used for myelodysplastic syndromes or acute promyelocytic leukemia, or biologically effective dose is reached. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. The biologically effective dose is defined as the dose at which 3 patients with constitutive STAT3 activity have the activity negated after the first dose of arsenic trioxide.

PROJECTED ACCRUAL: A maximum of 40 patients (6 for stratum I [accrued before November 2002] and 34 for stratum II [accrued since November 2002] will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed de novo or secondary acute myeloid leukemia with ≥ 20% blasts AND at least 1 of the following characteristics*:

  * Auer rods
  * Peroxidase or sudan black positive blasts
  * Chloroacetate esterase-positive or diffusely non-specific esterase-positive blasts
  * Presence of a myeloid immunophenotype by multiparameter flow cytometry, including expression of one or more myeloid markers (CD13, CD33) on blasts NOTE: *Megakaryocytic leukemia can be diagnosed by the detection of platelet antigens (e.g. factor VIII, glycoprotein Ib or IIb/IIIa) using monoclonal antibodies or the presence of ultrastructural platelet peroxidase
* No acute promyelocytic leukemia
* No Philadelphia-chromosome positive chronic myeloid leukemia
* Prior hematologic disorders, including myelodysplastic syndromes, aplastic anemia, paroxysmal nocturnal hemoglobinuria, and myeloproliferative disorders allowed

PATIENT CHARACTERISTICS:

Age

* 18 to 59

Performance status

* Not specified

Life expectancy

* More than 4 weeks

Hematopoietic

* Not specified

Hepatic

* Bilirubin ≤ 2 times normal*
* SGOT ≤ 2 times normal*
* Alkaline phosphatase ≤ 2 times normal* NOTE: *Unless abnormalities are directly attributable to leukemia

Renal

* Creatinine ≤ 1.5 times normal* NOTE: *Unless abnormalities are directly attributable to leukemia

Cardiovascular

* Cardiac ejection fraction ≥ 45%*
* Absolute QT interval ≤ 460 msec with potassium > 4.0 mEq/L and magnesium > 1.8 mg/dL
* No myocardial infarction within the past 6 months
* No uncontrolled symptomatic congestive heart failure
* No angina pectoris
* No multifocal cardiac arrythmias
* No other severe cardiovascular disease NOTE: *Unless abnormalities are directly attributable to leukemia

Other

* No serious medical or psychiatric illness that would preclude informed consent or limit survival to < 4 weeks
* No uncontrolled diabetes mellitus
* No other concurrent active malignancy
* No known hypersensitivity to E. coli-derived drug preparations
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for acute leukemia, except hydroxyurea to control white blood cell counts

  * Prior chemotherapy for an antecedent malignancy or other medical condition allowed

Endocrine therapy

* Not specified

Radiotherapy

* Prior radiotherapy for an antecedent malignancy or other medical condition allowed

Surgery

* Not specified

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2002-04; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and/or biologically effective dose or arsenic trioxide | 30 days after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Meir Wetzler, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States